CLINICAL TRIAL: NCT06446661
Title: Improving Oral Chemotherapy Adherence in Maintenance for Adolescents and Adults With Acute Lymphoblastic Leukemia Using Text Messages
Brief Title: Using Text Messages to Improve Oral Chemotherapy for Adolescents and Adults With Acute Lymphoblastic Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB23-1519
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Oral Chemotherapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity (Active Comparator): Receives high-intensity text messaging for 2 cycles of treatment
  Interventions: Other: High Intensity
- Low Intensity (Active Comparator): Receives no texts for 1st cycle and low-intensity texts for 2nd cycle
  Interventions: Other: No Text Messagings; Other: Low Intensity Text Messaging

INTERVENTIONS:
Other: High Intensity — Daily texts
  Arms: High Intensity
Other: No Text Messagings — Standard Care
  Arms: Low Intensity
Other: Low Intensity Text Messaging — Weekly Texts
  Arms: Low Intensity

SUMMARY:
The purpose of this section is to learn how text message reminders might help with regularly taking chemotherapy medications for Adolescents and Adults with Acute Lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
This study aims to compare adherence to oral mercaptopurine and methotrexate during the first 84-day cycle of maintenance therapy for adolescent and young adult patients with Acute Lymphoblastic Leukemia on pediatric-based regimens between those who receive the high intensity text message intervention and those who receive standard-of-care. It is believed that high-intensity text messages will increase patient adherence within cycle 1.

ELIGIBILITY:
Inclusion Criteria:

* Age of 15-39 years-old at the time of initial ALL diagnosis
* Diagnosed with ALL
* Currently receiving treatment with pediatric-based regimen that includes maintenance with mercaptopurine and methotrexate (e.g., CALGB 10403). Study participation begins with the start of maintenance, so enrollment occurs prior to the start of maintenance.

Exclusion Criteria:

* Patient or caregiver who would receive text message reminders does not have a cell phone that receives text messages
* Patient does not wish to participate
* Text messages will be crafted in the patient's preferred language for medical communication, so English fluency is not an enrollment requirement.

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
To compare adherence to oral chemotherapy with mercaptopurine and methotrexate | 84 days
  To compare adherence to oral mercaptopurine and methotrexate during the first 84-day cycle of maintenance therapy for patients with ALL on pediatric-based regimens between those who receive the high intensity text message intervention and those who receive standard of care.

SECONDARY OUTCOMES:
To describe the relationship between oral chemotherapy adherence and patient factors | 1 year
  At the start of cycle 1, Health Competence Beliefs Inventory (HCBI) scores will be collected as a baseline measurement of self-efficacy as measured in a prior AYA adherence study. Higher HCBI scores and lower ADI and SVM scores will be associated with higher adherence given prior associations with self-efficacy and family finances.

OTHER OUTCOMES:
To compare percentage of time during maintenance at goal absolute neutrophil count (ANC) and platelet count for patients | 1 year
  ANC and platelet measurements are collected throughout maintenance to monitor for therapeutic goals and the potential need for dose changes as part of AYA Oncology pharmacist-led management program
To compare clinical outcomes during and after maintenance therapy for AYA patients | 1 year
  Any changes in chemotherapy regimen or evidence of relapsed disease including new minimal residual disease (MRD) positivity within the first year of maintenance will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Study results including PHI such as dates, assigned study ID, and initials may be shared with researchers and their teams at other sites as part of required safety reporting notifications (e.g. serious events/unanticipated problems, or other reportable events). Final reports (no PHI) may also be shared. Names and medical record numbers will not be shared externally.
  Data will only be shared for analysis purposes.